CLINICAL TRIAL: NCT05291533
Title: Patient Experiences With Virtual Reality Mindfulness Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-06020347
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Distress, Emotional
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using VR Mindfulness Program (Other): Participants are inpatients on any NYP/WCM unit that use VR mindfulness programs; any patient referred for a psychological or neuropsychological evaluation by their treatment team will have the opportunity to complete the VR program. The study is seeking to evaluate the feasibility and preliminary efficacy of the VR mindfulness intervention.
  Interventions: Other: Virtual Reality (VR) Mindfulness Program

INTERVENTIONS:
Other: Virtual Reality (VR) Mindfulness Program — The VR program combines immersive, 3D visuals and audio with mindfulness skills practice. The program is designed to train participants you to calm their bodied and minds and its use is designed to enhance mindfulness practice. VR is a platform that has been used for a variety of applications, including gaming, entertainment, education and training.

SUMMARY:
This study aims to assess acceptability and preliminary efficacy of an intervention being administered clinically, a virtual reality (VR) mindfulness program. It is hypothesized that patients will find VR mindfulness an acceptable intervention and that it will reduce symptoms of anxiety.

DETAILED DESCRIPTION:
This pilot study proposes to assess acceptability and preliminary efficacy of an intervention being administered clinically, a virtual reality (VR) mindfulness program. Acceptability and preliminary efficacy will be determined by 1) patient feedback on their satisfaction with the intervention evaluated by the Client Satisfaction Questionnaire-8 (CSQ-8); 2) changes in acute subjective anxiety before and after using the program; 3) changes in subjective relaxation before and after using the program; 4) changes in global anxiety at referral to psychology and just prior to discharge; Any patient on units with access to this VR program who are referred for a psychological evaluation will have the opportunity to engage in the VR intervention.

Overall Design:

This study is an open trial evaluating the acceptability and efficacy of a VR mindfulness program being clinically implemented to address acute anxiety in patients admitted to medical and rehabilitation inpatient units.

VR Mindfulness Program:

Participants referred for a psychological or neuropsychological evaluation will have the opportunity to complete the study. A study staff member who is not the evaluating clinician will approach the patient to inquire about their interest in the study and conduct the informed consent process. Patients are typically referred for a psychological evaluation based on acute anxiety observed by staff or reported by the patient. The evaluating psychologist will collaborate with treatment team to make a clinical determination about whether VR mindfulness is indication (see exclusion criteria below). If it is determined that the patient could benefit from the VR intervention, a VR team member will facilitate the administration of a self-report measure on anxiety (GAD-7), obtain subjective ratings of anxiety and relaxation, and then administer the 5-minute VR mindfulness intervention. After patient's completion of the intervention, the VR team member will repeat the measures of subjective anxiety and relaxation. This procedure will be repeated as-needed (determined by clinical team) or up to three times per week based on patient preference and staff availability. The CSQ-8 will be administered after the patient's first use of VR mindfulness and again the day before discharge, if the patient opted to use repeatedly. The study team will re-administer the GAD-7 on the day prior to the patient's discharge.

Study-specific procedures:

Upon determination by the clinical and study team that a patient is an appropriate candidate for VR mindfulness, the patient will be informed of the opportunity to participate in the study. It will be made clear to the patient that participation in the study is voluntary and will have no impact on their current or future access to care at NYP/WCM. If they agree they will undergo the informed consent process.

Scientific Rationale for Study Design:

This is an open trial to determine acceptability and efficacy of using VR mindfulness to address acute anxiety in varied clinical settings. This intervention is already being implemented clinically, this study seeks to assess acceptability and provide preliminary data on efficacy of this intervention. No control is being used at this time.

4. Subject Selection

Subjects will be patients admitted to medical and rehabilitation inpatient units at NYP/WCM.

Recruitment:

Patients are identified by their clinical team during their inpatient admission as appropriate for the VR mindfulness intervention to address acute anxiety.

5. Registration Procedures

Subjects will be registered within the WRG-CT as per the standard operating procedure for Subject Registration.

6. Study Procedures Upon determination by the treatment team and VR team member that a patient is an appropriate candidate for VR mindfulness, the patient will be informed of the opportunity to participate in the study. It will be made clear to the patient that participation in the study is voluntary and will have no impact on their current or future access to care at NYP/WCM or their ability to participate in the VR mindfulness intervention. If they agree they will undergo the informed consent process.

Measures: Listed in the "Outcome Measures" section

Study intervention:

The study is seeking to evaluate the feasibility and preliminary efficacy of a VR mindfulness intervention. The VR program combines immersive, 3D visuals and audio with mindfulness skills practice. The program is designed to train participants you to calm their bodied and minds and its use is designed to enhance mindfulness practice. VR is a platform that has been used for a variety of applications, including gaming, entertainment, education and training.

Study duration, withdrawal and discontinuation:

Subjects will complete study procedures at least one time, with additional uses determined by need (decided by clinical team) or patient preference (up to three times per week based on staff availability). They will be followed for the duration of their admission. Study participation ends when they are discharged or are no longer eligible to use VR. Participants are free to withdraw from participation in the study at any time upon request.

An investigator may discontinue or withdraw a participant from the study for the following reasons:

* Significant study intervention non-compliance
* If any clinical adverse event (AE) or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the participant
* If the participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation
* Participant unable to participate in VR mindfulness intervention

The reason for participant discontinuation or withdrawal from the study will be recorded on the Case Report Form (CRF). Subjects who sign the informed consent form and do not receive the study intervention may be replaced. Subjects who sign the informed consent form and receive the study intervention, and subsequently withdraw, or are withdrawn or discontinued from the study will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Referred to psychology/neuropsychology
* Identified by treatment team for use of VR mindfulness intervention
* Able to provide informed consent or assent
* Patient is over the age of 18

Exclusion Criteria:

* Has not engaged in VR mindfulness intervention.
* Determination by clinical team that patient cannot or would not benefit from participation in VR.
* Reasons may include history of severe motion sickness or seizures, history of destruction of property, visual disturbance, vertigo, and cognitive impairment, delirium, and current or past diagnosis of a psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Change in composite score on Client Satisfaction Questionnaire-8 (CSQ-8; Attkisson & Zwick, 1982) | Immediately after first intervention (use of VR) and at hospital discharge an average of 10 days later
  An 8-item, empirically validated measure of satisfaction with a clinical program. Scores therefore range from 8 to 32, with lower values indicating lower satisfaction and higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
Mean change in Subject Units of Distress (SUDS) from pre- to post-VR | Immediately before and after each intervention (use of VR), up to two times per week for duration of hospital stay (average 10 days)
  This is a commonly used scale of 0 to 10 for measuring the subjective intensity of anxiety currently experienced by an individual. Scores range from 0 to 10, with lower values indicating lower distress and higher values indicating higher distress.
Mean change in Subjective units of relaxation from pre-to post-VR | Immediately before and after each intervention (use of VR), up to two times per week for duration of hospital stay (average 10 days)
  This scale is similar to SUDS, but asks patients to rate their subjective relaxation on a 0 to 10 scale. Scores range from 0 to 10, with lower values indicating lower relaxation and higher values indicating higher relaxation.
Mean change in General Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006) from baseline to discharge | Immediately before first intervention (use of VR) and at hospital discharge an average of 10 days later
  A 7-item, empirically validated, and gold-standard brief measure of global anxiety. Scores range from 0 to 21 with lower values indicating lower levels of anxiety and higher values indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Pelcovitz, Principal Investigator — Weill Cornell Psychiatry
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No